CLINICAL TRIAL: NCT00927095
Title: Continuous OC Treatment in PMDD: Steroid Hormone Mechanisms
Brief Title: Continuous Oral Contraceptive Treatment in Premenstrual Dysphoric Disorder (PMDD)
Acronym: PMDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Girdler, PhD, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH081837; R01MH081837 (NIH)
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Premenstrual Dysphoric Disorder
Keywords: PMDD; Oral contraceptives; steroid hormones; neurosteroids
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous OC (EE/DROS) (Active Comparator): Continuous daily oral drospirenone (DROS; 3mg) + ethinyl estradiol (EE; 20ug)
  Interventions: Drug: Continuous OC (EE/DROS)
- Intermittent OC (EE/DROS) (Active Comparator): Interrupted (21 days active - 7 days placebo) oral DROS (20ug)/EE(3mg)
  Interventions: Drug: Intermittent OC (EE/DROS)
- Placebo (Placebo Comparator): Continuous daily oral placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Continuous OC (EE/DROS) — Continuous EE(20ug)+DROS(3mg) daily for 3 months
  Other Names: Yaz
  Arms: Continuous OC (EE/DROS)
Drug: Intermittent OC (EE/DROS) — Intermittent EE(20ug)+DROS(3mg) daily for 21 days each month
  Other Names: Yaz
  Arms: Intermittent OC (EE/DROS)
Drug: placebo — daily placebo
  Other Names: oral placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare a low dose oral contraceptive (OC) given continuously (every day for three months) with the same low dose oral contraceptive given in an interrupted regimen (one week of inactive placebo pills each month) and with continuous placebo (inactive placebo given every day for three months). The primary hypothesis is that continuous OC will be significantly more effective in reducing premenstrual symptoms compared with either the interrupted OC or continuous placebo.

DETAILED DESCRIPTION:
Premenstrual Dysphoric Disorder (PMDD) describes the cyclic appearance of affective symptoms and resultant impairment during the luteal phase of the menstrual cycle. The objective of this trial is to determine if extended oral contraceptive (OC) regimens with eliminated pill-free intervals will successfully prevent the expression of PMDD symptoms. The central hypothesis of this application is that continuous administration of OCs will minimize the destabilizing effects of changing reproductive steroid levels and prevent PMDD symptom emergence. The cause of PMDD is unknown, the morbidity substantial, and the identified treatments limited in their effectiveness, since 40% of PMDD women are non-responders to elective serotonin re-uptake inhibitors (SSRIs). Earlier controlled studies of OCs to treat PMDD failed to find OCs superior to placebo using the traditional 21/7 platform (21 active pills followed by a 7 day pill-free interval (PFI)). Two recent trials of a low dose OC using a 24/4 platform did report greater reductions in premenstrual symptoms relative to placebo, presumably due to the shortened PFI. Despite the apparent efficacy of the 3-day extended dosing of this OC, the placebo response rate was substantial in these studies, resulting in a low effect size. Moreover, no steroid hormone levels were examined in these prior studies. In the absence of hormonal data, inferences about the mechanism of efficacy of extended OCs must remain speculative and untested.

Our proposed research will addresses the critical role of hormonal change in the precipitation of PMDD symptoms before and after treatment with a continuous OC regimen, an interrupted OC regimen (21/7 platform) and continuous placebo. This study will also permit us to examine the role of neurosteroids in PMDD. While acting acutely as anxiolytic positive modulators of the gamma-aminobutyric acid A (GABAA) receptor, these neurosteroids may paradoxically reduce the response of the GABAA receptor and cause irritability (in rats) following either extended exposure or withdrawal. Further, our prior research suggests that elevated levels of or changes in peripheral neurosteroid levels are associated with dysphoric mood symptoms in women with PMDD. Our hypothesis is that changes in neurosteroids modulate symptom severity rather than appearance in PMDD. The results of our study will suggest therapeutic targets and will inform future studies of both PMDD and related affective disorders.

ELIGIBILITY:
Inclusion Criteria:

* meets prospective criteria for PMDD, AND
* English speaking and reading skills.

Exclusion Criteria:

* current psychiatric disorder other than PMDD,
* history of venous thromboembolism,
* over 35 years of age and obese,
* uncontrolled hypertension or end-organ vascular disease,
* diabetes,
* migraine headache with aura,
* breastfeeding or pregnant,
* cigarette smoking,
* family history of premenopausal breast cancer or breast cancer in more than one first degree relative,
* elevated serum potassium levels, use of prescription medications (except stable thyroid supplementation),
* irregular menstrual cycles, OR
* history of: endometriosis, hepatic disease, breast carcinoma, pulmonary embolism or phlebothrombosis, malignant melanoma, cholecystitis or pancreatitis.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2008-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eisenlohr-Moul TA, Girdler SS, Johnson JL, Schmidt PJ, Rubinow DR. Treatment of premenstrual dysphoria with continuous versus intermittent dosing of oral contraceptives: Results of a three-arm randomized controlled trial. Depress Anxiety. 2017 Oct;34(10):908-917. doi: 10.1002/da.22673. Epub 2017 Jul 17. PMID 28715852

RESULTS

PARTICIPANT FLOW:
Groups:
- Continuous Low Dose Oral Contraceptive: continuous low dose oral contraceptive
  low dose oral contraceptive (20 ug ethinyl estradiol + 3 mg drospirenone): daily for three months
- Interrupted Low Dose Oral Contraceptive (21/7 Platform): interrupted low dose oral contraceptive (21/7 platform)
  20 ug ethinyl estradiol + 3 mg drospirenone: daily for 21 days each month
- Continuous Placebo: continuous placebo
  placebo: daily
Period: Overall Study
Arm/Group | Continuous Low Dose Oral Contraceptive | Interrupted Low Dose Oral Contraceptive (21/7 Platform) | Continuous Placebo
Started | 22 | 21 | 24
Completed | 16 | 17 | 22
Not Completed | 6 | 4 | 2
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Physician Decision | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Low Dose Oral Contraceptive | Interrupted Low Dose Oral Contraceptive (21/7 Platform) | Continuous Placebo | Total
Number analyzed (Participants) | 22 | 21 | 24 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (8.1) | 32.2 (8.6) | 32.1 (6.7) | 32.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 24 | 67
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 24 | 67

OUTCOME MEASURES:

1. Primary Outcome: Pre-Post Change in Premenstrual Symptom Severity
Description: Pre-post change (pre minus post) in mean premenstrual week severity of the worst emotional symptom as measured using the Daily Record of Severity of Problems items 1-8. Worst symptom for each individual was defined as the symptom in the baseline month demonstrating the highest mean severity during the premenstrual week. Mean premenstrual week severity scores were calculated to correspond to mean ratings; therefore, the mean premenstrual severity values ranged as follows: 1=Not at All, 2=Minimal, 3=Mild, 4=Moderate, 5=Severe, 6=Extreme. The change variable presented here is calculated as follows: "mean rating on the individual's worst symptom during the premenstrual week at baseline" minus "mean rating during the premenstrual week during the last on-treatment cycle". Therefore, higher values on this outcome variable correspond to greater reductions in premenstrual symptoms across the trial.
Time Frame: monthly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuous Low Dose Oral Contraceptive | Interrupted Low Dose Oral Contraceptive (21/7 Platform) | Continuous Placebo
Number analyzed (Participants) | 16 | 17 | 21
units on a scale | 1.93 (.22) | 1.73 (.22) | 1.64 (.19)

ADVERSE EVENTS:
Arm/Group | Continuous Low Dose Oral Contraceptive | Interrupted Low Dose Oral Contraceptive (21/7 Platform) | Continuous Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 22/22 | 21/21 | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Low Dose Oral Contraceptive (N=22) | Interrupted Low Dose Oral Contraceptive (21/7 Platform) (N=21) | Continuous Placebo (N=24)
Breast Tenderness (Reproductive system and breast disorders) | 15 (15) | 15 (15) | 18 (18)
Low Mood (Psychiatric disorders) | 17 (17) | 13 (13) | 17 (17)
Headache, Not Migraine (Nervous system disorders) | 10 (10) | 16 (16) | 20 (20)
Fatigue (General disorders) | 14 (14) | 17 (17) | 15 (15)
Irritability (Psychiatric disorders) | 14 (14) | 14 (14) | 15 (15)
GI Symptoms (Gastrointestinal disorders) | 13 (13) | 16 (16) | 13 (13)
Leg or Calf Discomfort (Musculoskeletal and connective tissue disorders) | 10 (10) | 13 (13) | 9 (9)
Anxious Symptoms (Psychiatric disorders) | 8 (8) | 8 (8) | 15 (15)
Bloating (Gastrointestinal disorders) | 4 (4) | 11 (11) | 10 (10)
Spotting (Reproductive system and breast disorders) | 11 (11) | 10 (10) | 4 (4)
Changing Bleeding Pattern - Prolonged Bleeding (Reproductive system and breast disorders) | 7 (7) | 4 (4) | 2 (2)
Headache, Migraine, No Aura (Nervous system disorders) | 5 (5) | 3 (3) | 3 (3)
Shortness of Breath or Chest Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Change in Bleeding Pattern (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 3 (3)
Suicidality (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Yeast Infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Heartburn or Reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache, Migraine, with Aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No